CLINICAL TRIAL: NCT03466164
Title: Neural Mechanisms of Mindfulness: a Discordant Twin Design
Brief Title: Neural Mechanisms of Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1R21AT009483 (NIH)
Record Dates: First submitted 2018-01-30; First posted 2018-03-15 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: discordant twin design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Mindfulness Based Stress Reduction Program (Experimental): Mindfulness-Based Stress Reduction MZ: identical (monozygotic; MZ) twins are tested in a pre-post manner, with only one twin randomly assigned to MT in between the two testing sessions
  Interventions: Behavioral: Mindfulness Based Stress Reduction Program
- Control MZ (No Intervention): Control MZ twin will complete 2 testing sessions without intervention.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Program — 8 week, 10-session course of mindfulness training
  Other Names: MBSR
  Arms: Behavioral: Mindfulness Based Stress Reduction Program

SUMMARY:
This project focuses on understanding the cognitive and neural mechanisms by which mindfulness training (MT) results in positive behavioral change and enhanced psychological well-being. Participants will complete two sets of cognitive tasks during functional magnetic resonance imaging (fMRI) and either be assigned to an MT intervention between scan sets or after scan sets.

DETAILED DESCRIPTION:
This project focuses on understanding the cognitive and neural mechanisms by which mindfulness training (MT) results in positive behavioral change and enhanced psychological well-being. Although MT is rapidly gaining in popularity as a life-style intervention, there are still critical gaps in our understanding of its primary mechanism of action. Current theoretical frameworks suggest that MT operates by improving attentional control, emotional regulation, and self-awareness capabilities, potentially by targeting neuroplastic brain mechanisms of executive control. This suggests an important role for cognitive neuroscience research, but current work is still in its infancy, and subject to a number of well-recognized methodological and conceptual limitations. The proposed project aims to systematically remedy these limitations of prior MT research, by leveraging the unique opportunities offered by the Human Connectome Project (HCP), and on-going NIH R01-funded research. A key feature of the project is the use of a randomized, longitudinal discordant twin design, in which monozygotic (MZ; identical) twin pairs will be recruited, with one co-twin randomly assigned to the MT condition (mindfulness-based stress reduction, or MBSR; the most-validated and standardized form of MT instruction) and the other serving as a (wait-list) control. Each co-twin will undergo extensive behavioral and MRI neuroimaging assessments in a pre/post fashion, before and after the MT (or no-contact control) intervention, to test for specific MT-related effects. The discordant twin design, though never previously employed in an MT context, is widely recognized as one of the strongest for causal inference, since it avoids many of the challenges and confounds associated with inadequately matched control groups, and enables twin-pair focused analyses, which greatly increase statistical power. The investigators will use this design to investigate theoretically-focused hypotheses that stem from a guiding framework regarding the neural mechanisms of cognitive control. Specifically, using a newly developed cognitive control task battery, the investigator will test the counter-intuitive hypothesis that MT produces an enhancement in the neural mechanism and circuits associated with reactive (rather than proactive) control. An additional subset of MZ twin participants will undergo retesting with the original HCP protocol, in order to provide a comprehensive assessment and comparison of MT effect sizes across multiple domains of cognitive and brain function. Success in this project will have high relevance for public health, by providing innovative experimental tools and a novel theoretical framework from which to empirically evaluate and better understand the potential impact of MT programs as lifestyle interventions for enhancing psychological well-being in healthy populations.

ELIGIBILITY:
Inclusion Criteria:

* monozygotic (MZ) or dizygotic (DZ) twins
* age range 22 to 45 years
* native English speaker

Exclusion Criteria:

* current psychiatric diagnosis
* taking psychoactive medication
* medical disorder that affects cognitive or motor function
* present or past head injury with documented neurological sequelae, and/or causing loss of consciousness.
* Pregnancy
* Claustrophobia
* Metallic objects
* Heart rhythm abnormalities or pacemaker
* Premature birth (before 34 weeks)

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in proactive cognitive control composite behavioral score | Baseline (0 months), Post (through study completion, an average of 3 months)
  The proactive composite variable consists aggregates the proactive condition of 4 tasks (Stroop, Cued Task-Switching, AX-CPT, Sternberg WM). For each task, a z-score is computed for each participant from their behavioral performance score: [(participant score - mean)/standard/deviation]. Then the composite score is created by summing z-scores.
Change in reactive cognitive control composite behavioral score | Baseline (0 months), Post (through study completion, an average of 3 months)
  The reactive composite variable consists aggregates the reactive condition of 4 tasks (Stroop, Cued Task-Switching, AX-CPT, Sternberg WM). For each task, a z-score is computed for each participant from their behavioral performance score : [(participant score - mean)/standard/deviation]. Then the composite score is created by summing z-scores.
Change in proactive cognitive control composite brain imaging activation score | Baseline (0 months), Post (through study completion, an average of 3 months)
  The proactive composite variable consists aggregates the proactive condition of 4 tasks (Stroop, Cued Task-Switching, AX-CPT, Sternberg WM). For each task, a z-score is computed for each participant from the brain activation score in the region of interest (ROI): [(participant score - mean)/standard/deviation]. Then the composite score is created by summing z-scores.
Change in reactive cognitive control composite brain imaging activation score | Baseline (0 months), Post (through study completion, an average of 3 months)
  The reactive composite variable consists aggregates the reactive condition of 4 tasks (Stroop, Cued Task-Switching, AX-CPT, Sternberg WM). For each task, a z-score is computed for each participant from the brain activation score in the region of interest (ROI): [(participant score - mean)/standard/deviation]. Then the composite score is created by summing z-scores.

SECONDARY OUTCOMES:
Psychological well-being | Baseline (0 months), Post (through study completion, an average of 3 months)
  Score on the Satisfaction with Life self-report measure
Mindfulness | Baseline (0 months), Post (through study completion, an average of 3 months)
  Score on the MAAS self-report measure
Anxiety | Baseline (0 months), Post (through study completion, an average of 3 months)
  Score on the STAI self-report measure
Positive and Negative Mood | Baseline (0 months), Post (through study completion, an average of 3 months)
  Score on the PANAS self-report measure

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT03466164/Prot_ICF_000.pdf